CLINICAL TRIAL: NCT04774185
Title: Hearing Aid Transmitter Performance Study - SRF-366
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-366
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2021-04

CONDITIONS: Hearing Loss
Keywords: Acoustical Coupling
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New hearing aid loudspeaker (Experimental): The new hearing aid loudspeaker is a loudspeaker system with a modified acoustic coupling approach which will be fitted based on the participants' individual ear anatomy.
  Interventions: Device: New hearing aid loudspeaker
- Standard hearing aid loudspeaker (Active Comparator): The hearing aid loudspeaker is a loudspeaker system with the existing acoustic coupling approach which will be fitted based on the participants' individual ear anatomy.
  Interventions: Device: Standard hearing aid loudspeaker

INTERVENTIONS:
Device: New hearing aid loudspeaker — The new hearing aid loudspeaker will be fitted to the participants individual ear anatomy and hearing loss.
  Arms: New hearing aid loudspeaker
Device: Standard hearing aid loudspeaker — The standard hearing aid loudspeaker will be fitted to the participants individual ear anatomy and hearing loss.
  Arms: Standard hearing aid loudspeaker

SUMMARY:
Sonova Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Sonova Hearing Systems undergo a final quality control in terms of clinical trials. This is a confirmatory study, investigating benefits of a modified hearing aid loudspeaker. This will be a clinical investigation which will be conducted mono centric at National Acoustic Laboratories a well known institution with exceptional experience (Australia).

DETAILED DESCRIPTION:
In this study a comparison with two Phonak Receiver in Canal (RIC) devices is done. The experimental device with a modified hearing aid loudspeaker concept and the active comparator with the existing technology will be compared regarding speech intelligibility, listening effort and sound quality in speech in noise, quiet situations for people with mild to moderate hearing losses.

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, mild to moderate Hearing loss)
* Good written and spoken English language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Willingness to wear Receiver in Canal hearing aids
* Informed Consent as documented by signature
* Normal cognitive abilities

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Sydney (AUS)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of speech intelligibility and sound quality for different loudspeaker | 2 weeks
  The Primary Outcome measure of this study is the comparison of the standard hearing aid loudspeaker with the modified one in regard to speech intelligibility in a noisy environment and sound quality in a quiet situation.
  The speech intelligibility will be measured using a speech test in dB SRT and the sound quality will be assessed by subjective rating, using percentage of satisfaction from "very satisfied (100)" to "very unsatisfied (0)".

SECONDARY OUTCOMES:
Evaluation of listening effort for different loudspeaker. | 2 weeks
  The Secondary Outcome measure of this study is the comparison of the standard hearing aid loudspeaker with the modified one in regard to listening effort in a noisy environment.
  The listening effort of speech will be assessed by subjective rating, within 13 steps, from "not effortful at all" to "only noise".
Evaluation of sound quality of own voice for different loudspeaker. | 2 weeks
  The Secondary Outcome measure of this study is the comparison of the standard hearing aid loudspeaker with the modified one in regard to sound quality in quiet.
  The sound quality of own voice will be assessed by subjective rating, using percentage of satisfaction from "very satisfied (100)" to "very unsatisfied (0)".
Evaluation of sound quality of streamed signals for different loudspeaker | 2 weeks
  The Secondary Outcome measure of this study is the comparison of the standard hearing aid loudspeaker with the modified one in regard to sound quality of a streamed signal in quiet and noise..
  The sound quality of the streamed signal will be assessed by subjective rating, using percentage of satisfaction from "very satisfied (100)" to "very unsatisfied (0)".

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Meijra, PhD, Principal Investigator — National Acoustic Laboratories
Locations (1):
- National Acoustic Laboratories, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ActiveVent™ Receiver provides benefit of open and --closed acoustics for better speech understanding in noise and naturalness of own voice perception — http://www.phonak.com/en-int/professionals/guides/evidence-library

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT04774185/Prot_SAP_000.pdf